CLINICAL TRIAL: NCT05906602
Title: Motor and Neurophysiological Changes After Ischemic Conditioning in Individuals With Stroke
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sangeetha Madhavan, Professor, Physical Therapy, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1620
Record Dates: First submitted 2023-02-17; First posted 2023-06-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to the type of ischemic conditioning they receive (real or sham). Treatment arms/ session order (ischemic conditioning and sham ischemic conditioning) will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ischemic Conditioning (Experimental): While seated, a rapid inflation cuff, similar to those used to measure blood pressure, will be placed around the paretic thigh to perform real ischemic conditioning. The pressure of the cuff will be increased for 5 minutes followed by no pressure for 5 minutes, repeated 5 times for a total of 50 minutes.
  Interventions: Device: Real Ischemic Conditioning
- Sham Ischemic Conditioning (Sham Comparator): While seated, a rapid inflation cuff, similar to those used to measure blood pressure, will be placed around the paretic thigh to perform sham or fake ischemic conditioning. The pressure of the cuff will be increased for 5 minutes followed by no pressure for 5 minutes, repeated 5 times for a total of 50 minutes.
  Interventions: Device: Sham Ischemic Conditioning

INTERVENTIONS:
Device: Real Ischemic Conditioning — 10-minute cycles of blood flow restriction (5 minutes) followed by blood flow release (5 minutes), repeated 5 times for a total of 50 minutes.
  Arms: Ischemic Conditioning
Device: Sham Ischemic Conditioning — Sham ischemic conditioning will mirror ischemic conditioning procedures, differing solely in cuff pressure during blood flow restriction to replicate to replicate perceived tightness without arterial blood flow restriction.
  Arms: Sham Ischemic Conditioning

SUMMARY:
The goal of this clinical trial is to test ischemic conditioning (blood flow restriction) as a neuromodulatory technique to improve gait function in stroke. Neuromodulation is emerging as a promising adjunct strategy to facilitate changes in brain activity and improve motor behavior following a neurological injury such as stroke.

The main questions this trial aims to answer are:

* Can ischemic conditioning produce neuromodulatory changes in the lower limb primary motor cortex?
* Can ischemic conditioning be used as a neuromodulatory technique to improve strength, motor control, and gait speed in individuals with stroke when compared to sham ischemic conditioning?

Participants will take part in two sessions of ischemic conditioning where a cuff (similar to ones that measure blood pressure) will be placed around the thigh and inflated to one of two blood flow restriction pressures (real or sham). Each participant will experience measures of brain activity and motor behavior testing before and after both sessions (ischemic conditioning and sham ischemic conditioning).

Researchers will investigate ischemic conditioning as neuromodulation modality in stroke to see if ischemic conditioning can produce beneficial changes in brain activity and improvements on subsequent motor behavior tasks.

ELIGIBILITY:
Inclusion Criteria:

* Single, stroke > 6 months since onset
* Residual hemiparetic gait deficits (e.g., abnormal gait pattern)

Exclusion Criteria:

* Lesions affecting the brainstem or cerebellum
* Other neurological disorders that may interfere with motor function
* Unhealed decubiti, persistent infections that may interfere with ability to perform test procedures
* Significant cognitive or communication impairment (Mini-Mental State Examination (MMSE<21)), which could impede the understanding of the purpose of procedures of the study
* Botulinum toxin (Botox) treatments to the lower limb within the past 6 months
* Pregnant women
* Contraindications to transcranial magnetic stimulation (TMS) or ischemic conditioning (IC) (Listed below)

TMS General Exclusion Criteria:

* Previous adverse reaction to TMS
* Skull abnormalities or fractures
* Concussion within the last 6 months
* Unexplained, recurring headaches
* Implanted cardiac pacemaker
* Metal implants in the head or face
* History of seizures or epilepsy
* Use of medications that could alter cortical excitability or increase risk of seizure (e.g., antidepressants, antipsychotics, anxiolytics, anticonvulsants)
* Current pregnancy

IC General Exclusion Criteria:

* History of thrombosis (i.e., blood clots) including venous thrombosis or deep vein thrombosis (DVT).
* Blood clots in the leg, or any condition in which compression of the thigh or transient ischemia is contraindicated (i.e., open wounds in the leg, bruising, nerve damage, etc.)
* Peripheral arterial grafts in the lower extremity
* History of uncontrolled hypertension
* History of peripheral vascular disease or hematological disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in corticomotor excitability | Changes in corticomotor excitability will be calculated within and between sessions at baseline, immediate-post, and 30-minutes-post one session of sham IC, real IC, and aerobic exercise.
  Excitability of the primary lower limb motor cortex will be assessed using single pulse transcranial magnetic stimulation (TMS) and motor evoked potentials (MEPs) will be recorded from the tibialis anterior muscle of the paretic leg.
Change in transcallosal inhibition | Changes in transcallosal inhibition will be calculated within and between sessions at baseline, immediate-post, and 30-minutes-post one session of sham IC, real IC, and aerobic exercise.
  Inhibition from the stimulated hemisphere to the non-stimulated hemisphere will be quantified as a measure of the ipsilateral silent period (iSP) using single pulse transcranial magnetic stimulation (TMS) and motor evoked potentials (MEPs) will be recorded from the tibialis anterior muscle of the leg ipsilateral to TMS stimulation.
Change in ankle motor control | Changes in ankle motor control will be calculated within and between sessions at baseline, immediate-post, and 30-minutes-post one session of sham IC, real IC, and aerobic exercise.
  Reaction time will be measured using a choice reaction time task involving rapid ankle dorsiflexion and plantarflexion movements in a custom built ankle-tracking device.
Change in lower limb strength | Changes in strength will be calculated within and between sessions at baseline, immediate-post, and 30-minutes-post one session of sham IC, real IC, and aerobic exercise.
  Participants will perform 3 trials each of maximum ankle dorsiflexion and plantarflexion strength.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) for Pain | During each real and sham ischemic conditioning session, pain scores will be reported for each participant during intervals of blow flow restriction and reperfusion through study completion, an average of 1 year.
  Subjective measures of pain will be reported during ischemic conditioning and sham ischemic conditioning using a Numerical Rating Scale (NRS) from 0 (no pain) to 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Madhavan, PT, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No